CLINICAL TRIAL: NCT00231517
Title: Randomised Double Blind Placebo Controlled Cross Over Design of the Efficacy of Topical Morphine for Inflammatory Pain in Children With Epidermolysis Bullosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01MH17
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2005-10

CONDITIONS: Epidermylosis Bullosa
MeSH Terms: interventions — Morphine; IntraSite Gel

INTERVENTIONS:
Drug: topical opiod
Drug: morphine sulphate in intrasite gel

SUMMARY:
Randomised Double blind placebo controlled cross over design study of the efficacy of morphine for inflammatory pain in children with Epidermolysis Bullosa

ELIGIBILITY:
Inclusion Criteria:

* children under 18 years epidermolysis wounds requiring dressing changes

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Richard Howard, Prof, Principal Investigator — Institute of Child Health
Locations (1):
- Great Ormond Street Hospital and the Institute of Child health, London, United Kingdom